CLINICAL TRIAL: NCT03622931
Title: Double-blind, Placebo-controlled Multicenter Phase II Trial to Evaluate the Efficacy and Safety of Romiplostim for the Treatment of Chemotherapy-induced Thrombocytopenia in Subjects With Relapsed Ovarian Cancer (2nd or Further Line)
Brief Title: Patients With Relapsed Ovarian Cancer (2nd and 3rd Line) Treated With Chemotherapy According to AGO Guidelines
Acronym: TRACEII
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to lack of recruitment
Sponsor: Gesellschaft fur Medizinische Innovation - Hamatologie und Onkologie mbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T-RACE II
Record Dates: First submitted 2018-01-18; First posted 2018-08-09 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Ovarian Cancer
Keywords: ovarian; cancer; romiplostim; nplate
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — romiplostim

STUDY DESIGN:
Intervention Model Description: 74 patients (about 37 in the experimental and 37 in the placebo arm), evaluable for the principal efficacy endpoint, are required. These will be recruited from an expected number of 15 sites.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- the experimental arm (Experimental): standard chemotherapy at 3/4-weekly intervals (cf. inclusion criteria) + romiplostim 750 μg sc once per week for up to 4 cycles
  Interventions: Drug: Standard chemotherapy; Drug: Romiplostim
- the placebo arm (Placebo Comparator): standard chemotherapy at 3/4-weekly intervals (cf. inclusion criteria) + placebo once per week for up to 4 cycles
  Interventions: Drug: Standard chemotherapy; Drug: Placebos

INTERVENTIONS:
Drug: Standard chemotherapy — Chemotherapy
Drug: Romiplostim
  Arms: the experimental arm
Drug: Placebos
  Arms: the placebo arm

SUMMARY:
To evaluate the safety of secondary chemotherapy induced thrombocytopenia (reduction in platelets which leads to bleeding) prophylaxis with romiplostim in ovarian cancer subjects receiving myelosuppressive (blood cell damaging) chemotherapy.It is anticipated that Romiplostim, when administered at an effective dose and schedule, will be a well-tolerated treatment for subjects experiencing chemotherapy-induced thrombocytopenia.

DETAILED DESCRIPTION:
Chemotherapy of recurrent ovarian cancer leads to severe thrombocytopenia in a considerable proportion of the patients, requiring treatment delays or dose reductions, and placing the patient at a high risk of bleeding complications. The amount of thrombocytopenia is highly schedule-dependent. In platinum-sensitive ovarian cancer that relapsed more than 6 months after end of primary therapy, a platinum containing reinduction therapy - the combination of paclitaxel/carboplatin, gemcitabine/carboplatin or PLD/carboplatin - is recommended according to the current AGO guidelines or recent ASCO presentations. Especially the latter two regimens often induce severe and even dose-limiting myelosuppression, including thrombocytopenia. Therefore, prophylaxis, or at least secondary prophylaxis of this toxicity is an important goal of supportive therapy. The use of platelet transfusions is limited by cost, supply problems, and associated risks, such as transfusion reactions, transmission of infection, and alloimmunization and platelet refractoriness. In contrast to the situation for the red and white blood cell compartments, the implementation of growth factor treatment in order to ameliorate the therapy of thrombocytopenia and its complications, is yet very limited. Romiplostim is an active second-generation thrombopoietic agent without safety problems due to immunogenicity, which proved to be beneficial in the treatment of immune thrombocytopenic purpura and myelodysplastic syndromes. The rationale of this trial is to obtain evidence that romiplostim can improve platelet counts/recovery in the treatment of recurrent ovarian cancer. Due to the fact, that the expected occurrence of severe thrombocytopenia and its complications may heavily depend on the selection of patient and their characteristics such as actually chosen treatment schedule, tumor stage, extent of metastasis, pre-treatment etc. a phase II design comparing the results to historical data or expectations is insufficient. A simple within-group control design, comparing subsequent cycles of the same patients with or without the supportive experimental drug may also be flawed, as "spontaneous" improvements after obviously unchanged chemotherapy are often observed. With some regimens, the first cycle proves to be generally more toxic than later ones. On the other hand, regimens may result in cumulative myelosuppression. A design including a randomized doubleblind control group is therefore warranted, moreover, as platelet counts represent a sensitive and valid surrogate marker for a clinical benefit. The current study will employ a model of secondary prophylaxis. The enrolment of subjects with grade 3 and/or 4 thrombocytopenia will facilitate an assessment of the ability of romiplostim to impact thrombocytopenia at clinically significant levels, which warrant the administration of platelet transfusions, dose reduction, and dose delay.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years of age
* Before any study-specific procedure, the appropriate written informed consent must be obtained, according to ICH-GCP, and national/local regulation
* ANC ≥ 1,000/μl, Hgb ≥ 9.5 g/dl, and platelet count ≥ 100 x 109/l on day 1 of the first on study cycle of the chemotherapy treatment (on-study cycle) (Thrombocytopenia have to be defined during a "qualifying cycle"; qualifying cycle could be the 1st or the 2nd cycle of the palliative chemotherapy; thrombocytopenia as evidenced by a platelet count < 50 x 109/l during the qualifying cycle of chemotherapy OR platelet count < 100 x 109/l on the planned starting day of the next cycle of chemotherapy (or 1-3 days before), requiring dose delay for platelet recovery.)
* Subjects with histologically confirmed advanced or metastatic ovarian cancer, fallopian tube cancer, peritoneal carcinoma or ovarian carcinosarcoma who are receiving 2nd or further line chemotherapy consisting of one of the following regimens according to established dosing standards:

  1. Topotecan, d 1-5, q3w
  2. Gemcitabine, d1+8, q3w
  3. Carboplatin / paclitaxel, d1, q3w
  4. Carboplatin d1 /gemcitabine, d1+d8, q3w
  5. Carboplatin / pegylated liposomal doxorubicin, d1, q4w
  6. Carboplatin d1 / gemcitabine, d1+d8, Avastin d1, q3w
  7. Topotecan d1-5 + avastin, q3w
  8. Carboplatin + paclitaxel + avastin, q3w
* Thrombocytopenia as evidenced by a platelet count < 50 x 109/l during the qualifying cycle of chemotherapy OR platelet count < 100 x 109/l on the planned starting day of the next cycle of chemotherapy (or 1-3 days before), requiring dose delay for platelet recovery; qualifying cycle could be the 1st or the 2nd cycle of chemotherapy
* Life expectancy ≥ 12 weeks at the time of screening
* Ability to receive the same dose and schedule of chemotherapy during the first on study treatment cycle as was given in the qualifying cycle(s). (In case of grade 4 thrombocytopenia: a dose reduction to ≥75% of the previous dose schedule is allowed.)

Exclusion Criteria:

* Previous treatment with PEG-rHuMGDF, recombinant human thrombopoietin (rHuTPO), romiplostim, eltrombopag, or another thrombopoietic protein
* Past or current history of malignancies that affect the overall prognosis (Please note: patients with past or current malignancies not affecting the overall prognosis are allowed for enrollment)
* Subjects, who have had a larger surgery within the last 2 weeks before entering this study
* Active participation in any other clinical study
* Subjects with an active infection; sepsis, disseminated intravascular coagulation, or any other condition (i.e. myelodysplastic syndrome {MDS}, immune thrombocytopenic purpura {ITP}, thrombotic thrombocytopenic purpura {TTP}, hemolytic uremic syndrome {HUS}) that may have exacerbated thrombocytopenia
* History of unstable angina, CHF {NYHA >class II}, uncontrolled hypertension {diastolic >100mm HG}, uncontrolled cardiac arrhythmia, or recent (within 1 year of screening) myocardial infarction (MI)
* History of arterial thrombosis (e.g., stroke or transient ischemic attack) within 1 year of screening
* History of pulmonary embolism or other venous thrombosis within 1 year of screening (except for catheter-related clots)
* Receipt of any experimental therapy within the last 4 weeks prior to screening; subject is currently enrolled in, or has completed within the last 30 days, another investigational device or drug study (exception: PROVE study)
* Receipt of a bone marrow or peripheral blood stem cell infusion (within 1 year of screening)
* Positive Pregnancy test
* breast feeding period
* Reproductive potential and not using adequate highly effective methods of contraceptive precautions in the judgment of the investigator during treatment and for 6 month (male or female) after the end of treatment (adequate: oral contraceptives, intrauterine device or barrier method in conjunction with spermicidial jelly)
* Known hypersensitivity to any recombinant E. Coli-derived product or any additives
* Inability to comply with the protocol or missing written informed consent
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the subject before registration in the trial.
* Accommodation in an institution due to official or legal orders (§40 p.1 No. 4 AMG)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Grade 3 and 4 thrombocytopenia | At the end of Cycle 1 (each cycle is 28 days)
  Platelet Count (100 x 10^9/L) will be measured and the rate will be compared by Treatment Group

SECONDARY OUTCOMES:
Adverse events of grade 3/4 | At the end of Cycle 4 (each cycle is 28 days)
  Determine the rate of AE between the experimental arm and the placebo arm.
Grade 3/4 thrombocytopenia | on days 8, 11 or 12, 15
  The rate of AE between the experimental arm and the placebo arm will be determined
Platelet Counts | on days 8, 11 or 12, 15
  The average platelet nadir in each treatment Group will be considered
Bleeding events | At the end of Cycle 8 (each cycle is 28 days)
  The proportion of patients suffering from grade 1, 2, 3, or 4 bleeding Events will be considered
Grade 1, 2, 3, or 4 thrombocytopenia (maximum NCI CTC grade by patient) | At the end of Cycle 8 (each cycle is 28 days)
  Determine the proportion of subjects in each treatment group
Grade 3/4 thrombocytopenia | At the end of Cycle 8 (each cycle is 28 days)
  The duration will be considered
Platelet transfusions | At the end of Cycle 8 (each cycle is 28 days)
  The number of subjects in each treatment Group will be considered
Platelet counts | On day 22 of each Cycle till max. 8 Cycles (each cycle is 28 days)
  The platelet counts on study chemotherapy treatment cycles by treatment group will be considered.
Counts of CT cycles | through study completion, an average of 8 month
  The proportion of subjects able to receive all CT cycles on time by treatment group
ADR/SADR of romiplostim | through study completion, an average of 8 month
  Assess the reported ADR/SADR

CONTACTS AND LOCATIONS:
Overall Officials: Jalid Sehouli, Prof. Dr. med., Principal Investigator — Frauenklinik
Locations (13):
- Germany (13):
  - Praxisklinik für Krebsheilkunde für Frauen Drs. Kittel /Klare / Wetzel, Berlin
  - Charité Campus Virchow-Klinikum Universitätsmedizin Berlin, Berlin
  - Ev. Waldkrankenhaus Spandau, Berlin
  - Gynäkologisches Zentrum, Bonn
  - Städtisches Klinikum Brandenburg, Brandenburg
  - Gemeinschaftspraxis Dr. Lorenz, Hecker, Wesche, Braunschweig
  - Klinikum Chemnitz GmbH, Chemnitz
  - Universitätsklinik Carl Gustav Carus der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Jena, Jena
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Caritasklinik St. Theresia Saarbrücken, Saarbrücken
  - Universitätsklinikum Tübingen, Tübingen